CLINICAL TRIAL: NCT01765400
Title: Platelet Reactivity With Clopidogrel Versus Prasugrel in Patients With Systolic Heart Failure
Brief Title: Platelet Inhibition in Patients With Systolic Heart Failure
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Daiichi Sankyo (Industry); Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 0574-11-FB
Record Dates: First submitted 2012-12-12; First posted 2013-01-10 (Estimated); Results first posted 2022-11-30 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-09

CONDITIONS: Systolic Heart Failure
Keywords: Heart failure; Antiplatelet therapy; Platelet aggregation; Clopidogrel; Prasugrel
MeSH Terms: conditions — Heart Failure, Systolic; Heart Failure | interventions — Prasugrel Hydrochloride; Clopidogrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prasugrel (Active Comparator): Prasugrel oral 10 mg once daily for 2 weeks
  Interventions: Drug: Prasugrel 10 mg daily x 2 weeks
- Clopidogrel (Active Comparator): Clopidogrel oral 75 mg once daily for 2 weeks
  Interventions: Drug: Clopidogrel 75 mg daily x 2 weeks

INTERVENTIONS:
Drug: Prasugrel 10 mg daily x 2 weeks
  Arms: Prasugrel
Drug: Clopidogrel 75 mg daily x 2 weeks
  Arms: Clopidogrel

SUMMARY:
The investigators aim to determine if patients with systolic heart failure treated with prasugrel achieve greater platelet inhibition compared to those treated with clopidogrel.

DETAILED DESCRIPTION:
Thienopyridine antiplatelet agents are an important component of therapy for management of acute coronary syndrome (ACS). Dual antiplatelet therapy with a thienopyridine, most commonly clopidogrel, and aspirin is widely used in the management of ACS to prevent major adverse cardiovascular events. Despite the benefits of this regimen, many patients continue to develop atherothrombotic events while on this regimen. Various reasons including inter-patient variability, delayed onset of action, and the obtainable antiplatelet activity of clopidogrel have been described as potential causes of the limited efficacy in preventing recurrent events. The Trial to assess improvement in therapeutic outcomes by optimizing platelet inhibition with prasugrel-thrombolysis in myocardial infarction (TRITON-TIMI 38) showed that patients with moderate-to-high-risk ACS scheduled for percutaneous coronary intervention (PCI) treated with prasugrel had decreased cardiovascular events compared to clopidogrel.

Clopidogrel is a prodrug that requires two hepatic conversion steps by the cytochrome (CYP)P450 enzyme system. The need for CYP450 involvement is known to contribute to the variable response of platelet inhibition demonstrated with clopidogrel. Although prasugrel is also a thienopyridine, it only requires hepatic CYP450 enzymes for one conversion step, and is converted to the active metabolite more efficiently. Therefore, prasugrel provides significantly more potent platelet inhibition compared to clopidogrel.

Patients with advanced systolic heart failure commonly have elevated hepatic venous pressures that can cause hepatic congestion and hypoperfusion resulting in impaired hepatic function. The elevated hepatic venous pressure predominantly affects the hepatic centrilobular cells which contain the highest concentration of cytochrome P-450 (CYP450) enzyme system. Hence patients with advanced heart failure may convert less clopidogrel to the active metabolite and subsequently produce less platelet inhibition compared to prasugrel.

Since prasugrel only requires the CYP450 system for one conversion step, the impact of hepatic congestion should be limited for heart failure patients treated with prasugrel. The phase 3, multi-center TRITON-TIMI 38 trial comparing clopidogrel and prasugrel showed that in an unselected patient population presenting with ACS, prasugrel achieved greater cardiovascular event reduction that was attributed to more robust platelet inhibition. Hence, we designed this trial to prospectively test the hypothesis that systolic heart failure patients with increased circulating catecholamines and possible abnormal functioning of CYP450 system treated with prasugrel will achieve greater platelet reactivity inhibition compared to those treated with clopidogrel.

ELIGIBILITY:
Inclusion Criteria:

* Patients 19 to 74 years of age.
* Patients with a left ventricular ejection fraction <35% by echocardiogram, SPECT myocardial perfusion study, cardiac MRI, cardiac computerized tomographic angiogram or invasive left ventricular angiogram within the last 6 months.
* Patients with NYHA Class III-IV heart failure at the time of enrollment.

Exclusion Criteria:

* Recent hospitalization within 30 days
* Patients expected to undergo major surgery or PCI in the next 30 days
* Patients taking clopidogrel, prasugrel, ticagrelor, ticlopidine, or cilostazol
* Patients listed for heart transplantation or having left ventricular assist device placement
* Patients with known allergy to either medication
* Patients with prior history of stroke or transient ischemic attack
* Patients with known intracranial neoplasm, aneurysm, or arteriovenous malformation
* Patients with a history of bleeding requiring hospitalization for treatment
* Patients taking oral anticoagulants
* Patients with body weight <60 kg
* Women who are pregnant or breastfeeding
* Patients with hemoglobin <10 mg/dl or platelet count <100,000/ul at baseline
* Patients with known clotting or platelet disorders
* Patients with a baseline INR > 1.4
* Patients with liver function tests (AST or ALT) > 2 times normal
* Patients with a suspected change in their use of aspirin during the study (starting, stopping, or changing dose of aspirin)
* Patients unwilling to consent to CYP2C19 genetic testing.

Ages: 19 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-05-15 (Actual); Primary Completion 2015-12-01 (Actual); Study Completion 2015-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Paul P Dobesh, PharmD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebaska Medical Center, Omaha, Nebraska, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Prasugrel: Prasugrel 10 mg once daily first for 14 days, then Clopidogrel 75 mg once daily for 14 days
- Clopidogrel: Clopidogrel 75 mg once daily first for 14 days, then Prasugrel 10 mg once daily for 14 days
Period: First Intervention (14 Days)
Arm/Group | Prasugrel | Clopidogrel
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0
Period: Second Intervention (14 Days)
Arm/Group | Prasugrel | Clopidogrel
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: 15 patients received prasugrel 10 mg once daily first for 14 days, then clopidogrel 75 mg once daily for 14 days 15 patients received clopidogrel 75 mg once daily first for 14 days, then prasugrel 10 mg once daily for 14 days
Groups:
- Prasugrel: Prasugrel 10 mg once daily for 2 weeks
  Prasugrel 10 mg daily x 2 weeks
- Clopidogrel: Clopidogrel 75 mg once daily for 2 weeks
  Clopidogrel 75 mg daily x 2 weeks
- Total: Total of all reporting groups
Arm/Group | Prasugrel | Clopidogrel | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 11 | 10 | 21
  >=65 years | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (8.9) | 58.5 (8.9) | 58.5 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 2 | 4
  White | 12 | 13 | 25
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: The Change in Platelet Aggregation Measured by the Accumetrics (VerifyNow P2Y12) Assay Between Baseline and Each Antiplatelet Medication
Time Frame: Baseline, 2 weeks post clopidogrel, and 2 weeks post prasugrel, Change From Baseline at Week 2 Reported
Measure: Mean (Standard Deviation); unit: PRU (P2Y12 reactivity units)
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 30 | 30
PRU (P2Y12 reactivity units) | 66.4 (51.5) | 156.2 (51.5)
Statistical Analysis 1: Comparison: Prasugrel; Test type: Superiority; p < 0.05, ANOVA

2. Secondary Outcome: The Change in Light Transmission Aggregometry (LTA)Between Baseline and Each Antiplatelet Medication
Time Frame: Baseline, 2 weeks post clopidogrel, and 2 weeks post prasugrel
Measure: Mean (Standard Deviation); unit: percentage of platelt inhibition
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 26 | 26
percentage of platelt inhibition
  5 umol/L ADP | 32 (18) | 47 (19)
  20 umol/L ADP | 38 (19) | 54 (18)

3. Secondary Outcome: The Change in Platelet Activation Assay (VASP)Between Baseline and Each Antiplatelet Medication
Time Frame: Baseline, 2 weeks post clopidogrel, and 2 weeks post prasugrel
Measure: Mean (Standard Deviation); unit: PRI (platelt reactivity index)
Arm/Group | Prasugrel | Clopidogrel
Number analyzed (Participants) | 26 | 26
PRI (platelt reactivity index) | 25 (20) | 49 (16)

ADVERSE EVENTS:
Arm/Group | Prasugrel | Clopidogrel
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 1/30 | 2/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prasugrel (N=30) | Clopidogrel (N=30)
Brusing (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No